CLINICAL TRIAL: NCT02411331
Title: Randomized, Multicenter, Double-blind, Vancomycin-controlled Study to Evaluate the Efficacy of Ethanol Lock Solution for the Curative Treatment of Implantable Venous Access Port Infection Due to Coagulase-negative Staphylococci
Acronym: Etha-LOCK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Centre Jean Perrin (Other); Jacques Lacarin Hospital Center (Other); CH Henri Mondor (Aurillac) (Unknown); Hôpital Nord (Saint-Etienne) (Unknown); University Hospital, Grenoble (Other); CH de Chambéry (Unknown); Hôpital de la Croix-Rousse (Other); Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-0232; 2014-A00488-39 (Registry Identifier: 2014-A00488-39)
Record Dates: First submitted 2015-04-03; First posted 2015-04-08 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Lock Solution; Catheter Related Blood Stream Infections; Central Venous Catheter Infection; Intravenous Drug Delivery Systems; Coagulase-negative Staphylococci Infection
Keywords: Lock Solution; Catheter related blood stream infections; Central venous catheter infection; Intravenous Drug Delivery Systems; Coagulase-negative staphylococci infection; Ethanol lock solution; Vancomycin lock solution
MeSH Terms: interventions — Ethanol; Enoxaparin; Vancomycin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Experimental group (Experimental): 90 patients will receive 10 injections of ethanol lock solution in implantable venous access port during the first 10 days of the study.
  Interventions: Drug: Ethanol 40% + Enoxaparine 400UI/ml
- control group (Other): 90 patients will receive 10 injections of vancomycin lock solution in implantable venous access port during the first 10 days of the study
  Interventions: Drug: Vancomycine 5 mg/ml + Héparine 2500UI/ml

INTERVENTIONS:
Drug: Ethanol 40% + Enoxaparine 400UI/ml
  Arms: Experimental group
Drug: Vancomycine 5 mg/ml + Héparine 2500UI/ml
  Arms: control group

SUMMARY:
Implantable venous access port infections are mainly due to coagulase negative staphylococci and may be managed by antibiotic lock therapy with retention of the port. Most of the time a vancomycin lock is used. Experimental data show that vancomycin may be poorly effective in eradicating the staphylococcal biofilm in the port. Another disadvantage of Vancomycin-containing lock solution is the occurrence of resistant organisms and the risk of catheter occlusion. Ethanol-containing lock solution is highly effective in vitro and does not expose to the risk of emergence resistance.

DETAILED DESCRIPTION:
Type of study: multi-center, randomized, double-blind, parallel-group, controlled clinical trial.

Number of centers: 9 French centers in Auvergne and Rhône-Alpes regions

Medical product Ethanol 40% + Enoxaparine 400UI/ml Versus Vancomycin 5 mg/ml + Héparine 2500UI/ml

Patients

Patients eligible for inclusion will be randomized to one of the two groups:

* Experimental group: 90 patients will receive 10 injections of ethanol lock solution in implantable venous access port during the first 10 days of the study.
* Control group: 90 patients will receive 10 injections of vancomycin lock solution in implantable venous access port during the first 10 days of the study.
* For each group, in case of bacteraemia, the lock therapy is associated with a systemic antibiotic therapy using another venous line and optimized by a specialist in infectious diseases.

Study Performance

Patients will be assessed at baseline D0, 3 days (D3), 10 days (D10), 14 weeks (W14) after D0 as follows:

Visit 1 (D0 - baseline):

* Signature of an informed consent form.
* Demographic and clinical characteristics (sex, age, disease associated with implantable venous access port, implantable venous access port infection data, bacteraemia data)

Days 1 to 10

* Injection of ethanol or vancomycin lock solution in implantable venous access port
* Ethanolemia 30 minutes after injection, on first day
* Side effects evaluation

Visit 2 (D3) and Visit 3 (D10)

* Side effects evaluation
* Blood culture
* Bacteraemia data (antibiotic therapy modification)

Phone contact each week from week 2 to week 13

End Visit (W14)

* Side effects evaluation
* Blood culture
* Bacteraemia data (antibiotic therapy modification)

ELIGIBILITY:
Inclusion Criteria:

* Man or woman from 18 years old
* With probable or definite implantable venous access port infection
* With or without bacteraemia
* Infection due to coagulase-negative staphylococci (except for lugdunensis Staphylococci)
* Blood culture results available within 48 hours before inclusion
* With health insurance

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Allergy to ethanol
* Patient with prosthetic cardiac valve
* Necessity of venous access port withdrawal
* Prior infection on the same venous access port
* Patients under supervision or (legal) guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Recovery at 12 week following the lock solution treatment completion | at 12 week
Favorable evolution without complication up to the end of implantable venous access port use | at 12 week
Favorable evolution without complication until the implantable venous access port withdrawal | at 12 week

SECONDARY OUTCOMES:
Negative peripheral and port blood cultures | at day 3 and day 10
Mortality due to infection of the port | at day 1
Implantable venous access port withdrawal rate | at day 1
Mechanical complication rate | at day 1
Blood alcohol concentration | 30 min after the first lock solution treatment
Side effects evaluation | at day 1

CONTACTS AND LOCATIONS:
Overall Officials: Olivier LESENS, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France